CLINICAL TRIAL: NCT02944227
Title: Efficacy of Fixed Monthly Dosing of Lucentis® (Ranibizumab) on Subretinal Fluid (SRF) Associated With Persistent Pigment Epithelial Detachment (PED) in Neovascular Age-related Macular Degeneration (AMD): A Pilot Study
Brief Title: Efficacy of Fixed Monthly Dosing of Ranibizumab in Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1512-107-728
Record Dates: First submitted 2016-02-16; First posted 2016-10-25 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Wet Macular Degeneration
MeSH Terms: conditions — Wet Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lucentis (Experimental): Lucentis fixed treatment
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: Lucentis — Lucentis fixed-treatment arm
  Other Names: Ranibizumab

SUMMARY:
The objective of this pilot study is to evaluate the efficacy of intensive fixed monthly dosing of intravitreal Lucentis® (Ranibizumab) for the treatment of SRF and PED in neovascular AMD which is persistent to anti-VEGF (anti-vascular endothelial growth factor) monotherapy.

DETAILED DESCRIPTION:
PEDs occur in up to 62% of eyes with advanced AMD. Numerous treatment options have been employed for PEDs in AMD, including laser therapies and intravitreal injections of anti-VEGF antibodies. However, eyes with PEDs were excluded from the larger clinical trials that used macular laser, photodynamic therapy, or ranibizumab to treat neovascular AMD; therefore, the efficacy of such options is still unclear for eyes with PEDs in neovascular AMD. Additionally, PED lesions have been reported to show less morphological and functional response to anti-VEGF monotherapy than eyes with other CNV lesions subtypes.

Based on the generally poor prognosis of PEDs and the lack of sufficient data in the literature regarding the effectiveness of fixed monthly dosing of Lucentis® (Ranibizumab) therapy, the investigators designed a prospective study to evaluate the effect of intensive fixed monthly dosing of Ranibizumab for the treatment of SRF associated with PED in neovascular AMD which is persistent to previous anti-VEGF monotherapy.

ELIGIBILITY:
Key inclusion criteria

1. Ability to provide written informed consent and comply with study assessments for the full duration of the study.
2. Age equal to or older than 50 years.
3. Presence of SRF associated with PED in neovascular AMD (proven with OCT FA, and ICG) which is persistent despite consecutive anti-VEGF injections for at least 9 months (3 initial loading doses with 4 week interval followed by PRN regimen)

   * A "persistent PED" is defined as a subject with < 50% reduction or increase in PED height

Key exclusion criteria

1. Administration of periocular, intravitreal, or systemic corticosteroid within 3 months prior to visit 1 in the study eye
2. Prior treatment with photodynamic therapy in the study eye
3. Previous subfoveal focal laser photocoagulation involving the foveal center in the study eye
4. Previous submacular surgery in the study eye
5. History of vitrectomy in the study eye
6. Epiretinal membranes (ERM)
7. Submacular hemorrhage or fibrosis within 50% of entire PED.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-08-21 (Actual)

PRIMARY OUTCOMES:
Changes of a pigment epithelial detachment (PED) | Baseline and 6 months
  Maximum height
Changes of a pigment epithelial detachment (PED) | Baseline and 6 months
  Maximum diameter
Changes of subretinal fluid (SRF) | Baseline and 6 months
  Maximum height
Changes of subretinal fluid (SRF) | Baseline and 6 months
  Maximum diameter

SECONDARY OUTCOMES:
Change in best corrected visual acuity from baseline | Baseline and 6 months
Changes in subfoveal thickness (SFT) measured by optical coherence tomography (OCT) from baseline | Baseline and 6 months
The proportion of cases maintaining vision and also who gained ≥ 15 letters from baseline | Baseline and 6 months
The proportion of cases having complete resolution of SRF associated with serous pigment epithelial detachment (PED) | Baseline and 6 months
The proportion of cases having complete resolution of subretinal fluid (SRF) associated with fibrovascular pigment epithelial detachment (PED) | Baseline and 6 months
The proportion of cases having persistent or recurrent subretinal fluid (SRF) associated with serous pigment epithelial detachment (PED) | Baseline and 6 months
The proportion of cases having persistent or recurrent subretinal fluid (SRF) associated with fibrovascular pigment epithelial detachment (PED) | Baseline and 6 months
The incidence of ocular adverse events | Through study completion, an average of 1 year
The proportion of cases experiencing leakage from neovascular AMD lesions | Baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chan CK, Abraham P, Sarraf D, Nuthi AS, Lin SG, McCannel CA. Earlier therapeutic effects associated with high dose (2.0 mg) Ranibizumab for treatment of vascularized pigment epithelial detachments in age-related macular degeneration. Eye (Lond). 2015 Jan;29(1):80-7. doi: 10.1038/eye.2014.233. Epub 2014 Oct 3. PMID 25277305
- [Background] Ersoy L, Ristau T, Kirchhof B, Liakopoulos S. Response to anti-VEGF therapy in patients with subretinal fluid and pigment epithelial detachment on spectral-domain optical coherence tomography. Graefes Arch Clin Exp Ophthalmol. 2014 Jun;252(6):889-97. doi: 10.1007/s00417-013-2519-9. Epub 2013 Nov 26. PMID 24271025
- [Background] Iordanous Y, Powell AM, Mao A, Hooper PL, Eng KT, Schwartz C, Kertes PJ, Sheidow TG. Intravitreal ranibizumab for the treatment of fibrovascular pigment epithelial detachment in age-related macular degeneration. Can J Ophthalmol. 2014 Aug;49(4):367-76. doi: 10.1016/j.jcjo.2014.05.010. PMID 25103655
- [Background] Arora S, McKibbin M. One-year outcome after intravitreal ranibizumab for large, serous pigment epithelial detachment secondary to age-related macular degeneration. Eye (Lond). 2011 Aug;25(8):1034-8. doi: 10.1038/eye.2011.115. Epub 2011 May 20. PMID 21597485